CLINICAL TRIAL: NCT05890495
Title: Patient-Applied Pretreatment Analgesia for Intrauterine Device Placement
Acronym: PAP-AID
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: American Academy of Family Physicians National Research Network (Network)
Responsible Party: Principal Investigator, Mike Arnold, Associate Professor, Uniformed Services University of the Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USUHS.2022-103
Record Dates: First submitted 2023-02-23; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Contraception
Keywords: Long-Acting Reversible Contraception
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Study medication provided per randomization table. Study participants allocated sequentially. Subject and provider blinded to allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Aqueous lidocaine (Experimental): Subject issued 5 ml jar of aqueous 4% lidocaine and will dip tampon distal end into jar for 30 seconds prior to placement.
  Interventions: Drug: Lidocaine topical; Device: Tampon
- Saline (Placebo Comparator): Subject issued 5 ml jar of sterile saline and will dip tampon distal end into jar for 30 seconds prior to placement.
  Interventions: Device: Tampon

INTERVENTIONS:
Drug: Lidocaine topical — 4% aqueous solution
  Other Names: Lidocaine hydrochloride topical solution, USP, 4%
  Arms: Aqueous lidocaine
Device: Tampon — Tampon with plastic applicator provided

SUMMARY:
The goal of this clinical trial is to perform a pilot study looking at the benefit of topical anesthetic application to the cervix by tampon prior to intra-uterine device insertion. The main question it aims to answer are:

* Does patient tampon-applied local anesthetic prior to insertion of an intrauterine device (IUD) reduce procedural duration?
* Does patient tampon-applied local anesthetic prior to insertion of an intrauterine device (IUD) reduce pain and improve patient perceptions of the procedure? Participants will place a tampon after dipping the tampon into the study-supplied medication (aqueous lidocaine or saline). Researchers will compare treatment and control groups to see if there is any difference in procedure time, difficulty or patient perceptions.

DETAILED DESCRIPTION:
This Pilot Randomized Double Blind Clinical Trial study will assess the effectiveness of patient-applied aqueous lidocaine via tampon as a pre-treatment prior to intra-uterine device placement. Subjects will apply the lidocaine or a saline placebo to the end of a standard tampon with a plastic applicator and then place the tampon 1 hour prior to the procedure. The tampon will be removed as the subject prepares for the procedure.

The procedure team will measure the procedure time as well as the subject and provider impressions of the procedure. This data will be evaluated to compare the lidocaine to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Request IUD insertion
* Age 18 or older
* Willingness to return for procedure after completing virtual study consent

Exclusion Criteria:

* Known allergy to viscous lidocaine or tampons
* Current vaginal or cervical injury

Ages: 18 Years to 54 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Procedure time | Measured during procedure
  Time from uterine sounding to cutting strings (to allow for procedures where an IUD is removed prior to placing a new IUD)
Patient-reported pain level | Obtained immediately after the procedure prior to the patient leaving the clinic
  0-10 Visual analog scale

SECONDARY OUTCOMES:
Patient-reported satisfaction with procedure | Obtained immediately after the procedure prior to the patient leaving the clinic
  0 - 100%
Patient-reported interest in subsequent procedure | Obtained immediately after the procedure prior to the patient leaving the clinic
  Likert scale
Provider-reported procedural difficulty | Obtained immediately after the procedure prior to the patient leaving the clinic
  Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Arnold, MD, Principal Investigator — Associate Professor, Uniformed Services University of the Health Sciences
Locations (1):
- University Family Health Center, USUHS, Bethesda, Maryland, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/95/NCT05890495/ICF_000.pdf